CLINICAL TRIAL: NCT00287417
Title: Nuchal Translucency Study - PAPP-A
Brief Title: Early Ultrasound and Maternal Biochemical Markers to Evaluate the Risk of Down Syndrome During the First Trimester
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Emmanuel LAVOUE, Directeur Adjoint de la DRCI, University Hospital, Strasbourg, France
Other Study IDs: 3032
Record Dates: First submitted 2005-09-13; First posted 2006-02-06 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Down Syndrome
Keywords: Nucal translucency; Down syndrome; MSS; Risk assessment
MeSH Terms: conditions — Down Syndrome | interventions — Ultrasonography; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Device: echography
Other: blood sample

SUMMARY:
The aim of the study is to evaluate the risk of Down syndrome during the first trimester of the pregnancy. The risk assessment is evaluated using early ultrasound and maternal biochemical markers.

ELIGIBILITY:
Inclusion Criteria:

* Female > 18 years old
* Pregnant

Exclusion Criteria:

* Maternal age < 18 years old, twin pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinics, public hospitals
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Actual)
Dates: Start 2003-07; Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Israel Nisand, MD, Principal Investigator — Hopitaux Universitaires de Strasbourg
Locations (7):
- France (7):
  - Département de Gynécologie-Obstétrique, Hôpital de Hautepierre, Hôpitaux Universitaires de Strasbourg, Strasbourg, Alsace
  - Service de Gynécologie-Obstétrique, SIHCUS, CMCO, Strasbourg, Alsace
  - Centre Hospitalier, Belfort
  - Centre Mère et Enfant LE PARC, Service de Gynécologie Obstétrique, Colmar
  - Centre de Périnatalité, Hôpital Civil, Guebwiller
  - Centre Hospitalier du Hasenrain, Mulhouse
  - Clinique ADASSA, Strasbourg